CLINICAL TRIAL: NCT06990204
Title: A Single Center, Open Label, Randomized, Four-period, Two-sequence, Fully Replicate, Cross-over Bioequivalence Study of Azilsartan Medoxomil 80 mg Tablets and Edarbi® 80 mg Tablets in Healthy Adult Subjects of Both Sexes Under Fasting Conditions
Brief Title: Bioequivalence Study of Azilsartan Medoxomil 80 mg Tablets (Gedeon Richter Plc., Hungary) and Edarbi® 80 mg Tablets (JSC Nizhpharm, Russia)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gedeon Richter Plc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EAEU-GCO-AZL-01-2024
Record Dates: First submitted 2025-04-28; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Hypertension
Keywords: Hypertension; High Blood Pressure; Azilsartan
MeSH Terms: conditions — Hypertension | interventions — azilsartan medoxomil; Tablets; azilsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azilsartan medoxomil 80 mg tablets (Experimental): 1 Azilsartan medoxomil 80 mg tablet (85.36 mg Azilsartan medoxomil potassium (Azilsartan Kamedoxomil) equivalent to 80 mg Azilsartan medoxomil)
  Interventions: Drug: Azilsartan medoxomil 80 mg tablet
- Edarbi® 80 mg tablets (Active Comparator): 1 Edarbi® 80 mg tablet (85.36 mg Azilsartan medoxomil potassium (Azilsartan Kamedoxomil) equivalent to 80 mg Azilsartan medoxomil)
  Interventions: Drug: Edarbi® 80 mg tablets

INTERVENTIONS:
Drug: Azilsartan medoxomil 80 mg tablet — 1 tablet of 80 mg of azilsartan medoxomil
  Arms: Azilsartan medoxomil 80 mg tablets
Drug: Edarbi® 80 mg tablets — 1 tablet of 80 mg of azilsartan medoxomil.
  Arms: Edarbi® 80 mg tablets

SUMMARY:
ACEis are among the most widely used classes of antihypertensive drugs. ARBs have a similar antihypertensive efficacy and protective effect as ACEis, albeit with a somewhat different mechanism for RAS inhibition and a smaller randomized clinical trials' database. A difference between ACEis and ARBs is their tolerability profile, with ARBs having a rate of side effects similar to placebo. Most importantly, the clinical evidence supports a relevant protective role of ARBs toward the CV and renal damage development, as well as the occurrence of major adverse CV events, in hypertensive patients. Moreover, a neutral metabolic effect has been reported upon ARBs administration, in contrast to other antihypertensive agents, such as BBs and diuretics. These properties highlight the use of ARBs as an excellent pharmacological strategy to manage hypertension and its dangerous consequences

The purpose of this study is to compare pharmacokinetics (PK), safety, and tolerability of the IMPs Azilsartan medoxomil 80 mg tablets and of Edarbi® 80 mg tablets in healthy adult subjects of both sexes under fasting conditions.

Dose proportionality in exposure was established for azilsartan in the azilsartan medoxomil dose range of 20 mg to 320 mg after single or multiple dosing. In the present study the highest available strength of Azilsartan medoxomil 80 mg tablets will be investigated. Administration of this dose is expected to provide accurate and reliable determination of azilsartan plasma concentrations.

This is a single center, open label, randomized, four-period, two-sequence, fully replicate, cross-over bioequivalence study in healthy adult subjects of both sexes after single dose administration under fasting conditions. A single oral dose of the IMP (Test IMP: Azilsartan Medoxomil 80 mg tablets or Reference IMP: Edarbi® 80 mg tablets )will be administered under fasting conditions in each of the 4 study periods.

ELIGIBILITY:
Inclusion Criteria:

1. Male or nonpregnant, nonlactating female volunteers, assessed as healthy by the Investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, vital signs (blood pressure, pulse rate, respiratory rate, body temperature) assessment, laboratory tests results (clinical chemistry, hematology, serology, and urinalysis), and cardiac monitoring (12-lead ECG).
2. Capable of voluntary, non-coerced provision of signed and dated informed consent form (ICF) prior to any study-specific procedures, which includes compliance with the requirements and restrictions listed in the ICF.
3. Aged 18-45 years inclusive at the time of signing the ICF.
4. Non-smokers (last episode of smoking or last use of tobacco- or nicotine-containing products more than 6 months prior to Screening, if any).
5. Body Mass Index (BMI) 18,5-30 kg/m2 inclusive and weight ≥50 kg and ≤ 120kg.
6. A valid (performed in accordance with the Clinical investigational site's standard operating procedures [SOPs]) negative SARS CoV 2 test result at Screening and upon each admission to the clinical unit.
7. Male volunteers (with the exception of vasectomised males) must be willing and able to use one of the following adequate methods of contraception from the first administration of the IMP until at least 30 days after the last administration of the IMP:

   * abstinence from penile-vaginal intercourse;
   * barrier contraception, i.e., a male condom plus spermicide (foam, gel, cream) when having penile-vaginal intercourse with a woman of childbearing potential.
8. Male volunteers must be willing to refrain from donating sperm from the first administration of the IMP until at least 30 days after the last administration of the IMP.
9. Female volunteers of childbearing potential (a woman is considered fertile following menarche and until becoming postmenopausal unless permanently sterile) who are using one of the adequate methods of contraception listed below consistently and correctly, must be willing and able to continue the use of the chosen adequate birth control method from 28 days prior to the first administration of the IMP until 28 days or 5 half-lives, whichever takes longer, after the last administration of the IMP in this study:

   * barrier contraception i.e., a male condom or female cervical cap plus spermicide (foam, gel, cream);
   * vasectomised partner;
   * abstinence from penile-vaginal intercourse;
   * bilateral tubal occlusion;
   * non-hormonal intrauterine device (IUD).
10. Female volunteers of non-childbearing potential, defined as:

    * postmenopausal (history of amenorrhea for ≥52 weeks without an alternative medical cause and confirmation by follicle-stimulating hormone (FSH) level consistent with post-menopause) or
    * surgically sterile (documented hysterectomy and/or bilateral salpingectomy and/or bilateral oophorectomy).

Exclusion Criteria:

1. History of, or ongoing allergy/hypersensitivity to any of the study IMPs, or components thereof, or drug or any other allergy.
2. Known history or presence of malignant disease.
3. History or presence of angioedema, cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, neuromuscular, psychiatric, auto-immune, or neurological disorders; history or presence of cerebrovascular diseases (including cerebral circulation failure), or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
4. Conditions associated with circulating blood volume decrease (including vomiting and diarrhea).
5. Any abnormalities in laboratory or instrumental test results which are outside the reference range of the Clinical investigational site.
6. Creatinine clearance <80 mL/min based on the Cockcroft-Gault equation.
7. Systolic blood pressure < 100 mmHg or > 130 mmHg; diastolic blood pressure < 70 mmHg or > 90 mmHg; pulse < 60 bpm or > 90 bpm.
8. Medical history of surgery on gastrointestinal tract and hepatobiliary system (excluding appendectomy).
9. Adherence to special types of diets (such as vegetarian, vegan, with salt restriction within 30 days prior to the first administration of the IMP) and lifestyle (work at night, extreme physical activity).
10. Difficulty fasting or consuming standard meals.
11. No suitable veins for cannulation or repeated venepuncture.
12. Any other condition that is capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the IMP; or interfering with the interpretation of data, as judged by the Investigator.
13. Use of any prescribed or nonprescribed medication including herbal remedies, vitamins, and minerals within 14 days prior to the first administration of the IMP or longer if the medication has a long half-life.
14. Use of drugs interacting with the IMP (for detailed list of concerned drugs, see Section 8.3.4) within 30 days prior to the first administration of the IMP.
15. Females who:

    * have used implanted, injected, intravaginal, or intrauterine hormonal contraceptives within 6 months prior to Screening;
    * have used oral or transdermal hormonal contraceptives within 1 month prior to Screening.
16. Have had a tattoo or body piercing within 30 days prior to the first administration of the IMP.
17. Presence of Hepatitis B surface antigen (HbsAg) at Screening or a Positive Hepatitis C antibody test (Anti-HCV) result at Screening.
18. Positive human immunodeficiency virus (HIV) antibody test result at Screening.
19. Positive Rapid Plasma Reagin (RPR or Treponema pallidum antibody) test result at Screening.
20. Volunteer was in contact with the person who had a positive test result for COVID 19 within 14 days prior to Screening.
21. Presence of one or more of the following signs/symptoms at any time during the study: cough, sore throat, shortness of breath or difficulty breathing at rest or with activity, body pain or muscle pain/aches, fatigue, headache, fever or chills, nasal obstruction or congestion, nasal discharge, nausea or vomiting, diarrhea, new loss of taste or smell, if confirmed by positive SARS CoV 2 test (rapid test) result.
22. Known or suspected history of drug abuse as judged by the Investigator.
23. Positive screen for drugs of abuse (to include at minimum: amphetamine, methamphetamines, cannabis, cocaine, opiates, barbiturates, benzodiazepine, methadone, tricyclic antidepressants) or alcohol at Screening or at any of the admissions to the clinical unit.
24. Positive urinary cotinine test at Screening or at any of the admissions to the clinical unit.
25. Regular alcohol consumption within 6 months prior to Screening, defined as an average weekly intake of >5 units of alcohol. One unit of alcohol is equivalent to: 500 mL of beer, 200 mL of dry wine or 50 mL of spirits.
26. Consumption of food containing poppy seeds within 72 h prior to Screening.
27. Any intake of red wine, Seville oranges, grapefruit or grapefruit juice, pomelos, exotic citrus fruits, grapefruit hybrids, or their juices within 7 days prior to the first administration of the IMP until collection of the final PK sample in this study.
28. Any intake of caffeine- or xanthine-containing products (e.g., coffee, tea, cola drinks, guaraná drinks, chocolate) within 48 h prior to the administration of the IMP until collection of the final PK sample during each dosing session.
29. Any intake of alcohol within 48 h prior to the administration of the IMP until collection of the final PK sample during each dosing session.
30. Participation in strenuous exercise within 48 h prior to the administration of the IMP until collection of the final PK sample during each dosing session.
31. Plasma donation within one month of Screening or any blood donation/blood loss >500 mL during the 3 months prior to Screening or ≥50 mL and <500 mL within 30 days prior to the first administration of the IMP.
32. The subject has participated in a clinical trial and has received an IMP within the following time period prior to the first administration of the IMP in the present study: 30 days, 5 half-lives or twice the duration of the biological effect of the IMP (whichever is longer), or recent participation in a clinical investigation that, in the opinion of the Investigator, would jeopardize subject's safety or the integrity of the study results.
33. Previous randomization to the IMP in the present study.
34. Known or ongoing psychiatric disorders that would interfere with study participation as determined by the Investigator.
35. Volunteer reports difficulty swallowing tablets whole.
36. Judgment by the Investigator that the healthy volunteer should not participate in the study if they are considered unlikely to comply with study procedures, restrictions, and requirements.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-06-06 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Bioequivalence of Azilsartan medoxomil 80 mg tablets and Edarbi® 80 mg tablets by measuring the AUC from time 0 to last collection time t (AUC0-t) | The duration of sampling period of 72 hours is sufficient to adequately describe the plasma concentration-time profile of azilsartan. The expected total study duration for each subject will be 26-42 days (considering 1-7 days for Screening).
  The primary purpose of the study is to assess the bioequiavelence of Azilsartan medoxomil 80 mg tablets (Gedeon Richter Plc., Hungary) and Edarbi® 80 mg tablets (JSC Nizhpharm, Russia) in healthy adult subjects of both sexes under fasting conditions. The 90% CI for the ratio of geometric means (T/R) based on least-squares means from the ANOVA of the ln-transformed AUC0-t for azilsartan must be within 80.00% to 125.00%.
Bioequivalence of Azilsartan medoxomil 80 mg tablets and Edarbi® 80 mg tablets by measuring the maximum concentration in plasma (Cmax) | The duration of sampling period of 72 hours is sufficient to adequately describe the plasma concentration-time profile of azilsartan. The expected total study duration for each subject will be 26-42 days (considering 1-7 days for Screening).
  The primary purpose of the study is to assess the bioequiavelence of Azilsartan medoxomil 80 mg tablets (Gedeon Richter Plc., Hungary) and Edarbi® 80 mg tablets (JSC Nizhpharm, Russia) in healthy adult subjects of both sexes under fasting conditions. 90% CI for the ratio of geometric means (T/R) based on least-squares means from the ANOVA of the ln-transformed Cmax must be within 80.00% to 125.00%.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From enrollment up to 6 weeks.
  The secondary purpose is to assess the safety and tolerability of the study products from the signing of the informed consent form (ICF) until the end of the study. There will be no formal statistical evaluation of safety or tolerability. The safety results will be provided as listings and summary tables for each treatment group. Adverse event data listing will include AEs onset and resolution date/time, duration, time from dosing, severity, relationship to the IMP and/or the additional drug product, outcome, and the action taken to the IMP and/or additional drug product and to treat the AE.

CONTACTS AND LOCATIONS:
Locations (1):
- LLC Professorskaya klinika, Perm, Perm Krai, Russia